CLINICAL TRIAL: NCT06166147
Title: A Proof of Concept Study of Pancreatic Cancer Early Detection by cfDNA Assay
Brief Title: A Prospective Study of Liquid Biopsy for Pancreatic Cancer Early Detection
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Collaborators: Shanghai Weihe Medical Laboratory Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xian-Jun Yu, Principal Investigator, Fudan University
Other Study IDs: Profound-PC
Record Dates: First submitted 2023-11-07; First posted 2023-12-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer arm: Participants with new diagnosis of pancreatic cancer, from whom a peripheral blood sample will be collected.
- Benign disease arm: Participants with benign pancreatic diseases, from whom a peripheral blood sample will be collected.

SUMMARY:
This study is a multi-center, observational study aiming at developing a machine learning-based early detection model using prospectively collected liquid biopsy samples from clinically-annotated individuals.

DETAILED DESCRIPTION:
Peripheral blood samples from participants with new diagnosis of pancreatic cancers will be collected to characterize the cancer-specific circulating signals by sequencing cell free DNA. A noninvasive test integrating machine learning algorithm will be trained and validated through a two-stage approach in recruited well-classified individuals, along with non-cancers without clinical diagnosis of cancer after routine medical screening. The performance of liquid biospy assays discovering cancer from non-cancer will be evaluated in participants with benign disease as well as average risk individuals.

ELIGIBILITY:
Cancer Arm

Inclusion Criteria:

* 40-75 years old
* Clinically and/or pathologically diagnosed pancreatic cancer
* No prior or undergoing any systemic or local antitumor therapy, including but not limited to surgical resection, radiochemotherapy, endocrinotherapy, targeted therapy, immunotherapy, interventional therapy, etc.
* Able to provide a written informed consent and willing to comply with all part of the protocol procedures.

Exclusion Criteria:

* Pregnancy or lactating women
* Known prior or current diagnosis of other types of malignancies comorbidities
* Severe acute infection (e.g. severe or critical COVID-19, sepsis, etc.) or febrile illness (body temperature of ≥ 38.0 °C) within 14 days prior to blood draw
* Recipients of organ transplant or prior bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 30 days prior to study blood draw
* Recipients of therapy in past 14 days prior to blood draw, including oral or IV antibiotics, glucocorticoid, azacitidine, decitabine, procainamine, hydrazine, arsenic trioxide
* Other conditions that the investigators considered are not suitable for the enrollment

Benign Disease Arm

Inclusion Criteria:

* 40-75 years old
* Clinically and/or pathologically diagnosed pancreatic non-malignant disease (pancreatic intraepithelial neoplasia, pancreatic cyst and chronic pancreatitis)
* No prior or undergoing any systemic or local antitumor therapy, including but not limited to surgical resection, radiochemotherapy, endocrinotherapy, targeted therapy, immunotherapy, interventional therapy, etc.
* Able to provide a written informed consent and willing to comply with all part of the protocol procedures

Exclusion Criteria:

* Pregnancy or lactating women
* Known prior or current diagnosis of other types of malignancies comorbidities
* Severe acute infection (e.g. severe or critical COVID-19, sepsis, etc.) or febrile illness (body temperature of ≥ 38.0 °C) within 14 days prior to blood draw
* Recipients of organ transplant or prior bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 30 days prior to study blood draw
* Recipients of therapy in past 14 days prior to blood draw, including oral or IV antibiotics, glucocorticoid, azacitidine, decitabine, procainamine, hydrazine, arsenic trioxide
* Other conditions that the investigators considered are not suitable for the enrollment

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed pancreatic cancer or pancreatic non-malignant disease
Sampling Method: Non-Probability Sample
Enrollment: 276 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Performance of cfDNA methylation-based model for discriminating pancreatic cancer versus non-cancer | 12 months
  Sensitivities of cfDNA methylation-based model at specificity of 99% and 95%, respectively.

SECONDARY OUTCOMES:
Performance of models using multi-omic data for discriminating pancreatic cancer versus non-cancer | 12 months
  Sensitivities of model integrating multi-omics data at specificity of 99% and 95%,respectively.
Performance of pre-defined model in clinical sub-groups of interest | 12 months
  Sensitivity of pre-defined model in different pathological subtypes or different age groups or tumor marker-negative cases.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Jun Yu, M.D., Ph.D., Study Chair — Fudan University
Locations (3):
- China (3):
  - Department of Pancreatic and Hepatobiliary Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality
  - Department of Hepato-Biliary-Pancreatic-Splenic Surgery, Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Department of General Sugery, Huadong Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No